CLINICAL TRIAL: NCT05425810
Title: R21: An Easy-to-use, iNtelligent, Affordable LinEr (ENABLE) System for Socket Fit Assessment
Acronym: ENABLE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: North Carolina State University (Other)
Responsible Party: Principal Investigator, Ming Liu, Research Assistant Professor, North Carolina State University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 23949
Record Dates: First submitted 2022-05-09; First posted 2022-06-21 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Lower Limb Amputation Below Knee (Injury)
Keywords: amputee; prosthetic socket; residual skin; pressure ulcer
MeSH Terms: conditions — Wounds and Injuries; Pressure Ulcer

STUDY DESIGN:
Intervention Model Description: All the participants will go through the same testing procedure. Both the experimenters and the participants know very well about the change in the experimental setup.
Masking Description: When the digital photos are shown to evaluators from external groups, the socket fitting conditions are not disclosed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Transtibial patient (Experimental): All the recruited participants will be included in this arm and will go through the socket manufacturing, fitting, and testing procedure.
  Interventions: Device: Apply ENABLE sensing pad; Device: Insert small pads at pressure tolerant locations

INTERVENTIONS:
Device: Apply ENABLE sensing pad — The developed ENABLE system is integrated into the standard prosthetic liner and measures the pressure distribution during locomotion. Using the ENABLE system may lead temporary increase in the temperature inside the prosthetic socket and it is expected that the total exposition during the experimental procedure will be less than 10 min.
Device: Insert small pads at pressure tolerant locations — To change the pressure distribution inside the socket, four fitting conditions are introduced by adding small pads at patella tendon (PT), lateral tibial crest (LTC), medial tibial crest (MTC), and popliteal fossa (PF) respectively. Including the no pads scenario, totally of five fitting conditions are simulated.

SUMMARY:
Lower limb amputees (LLA) rely on their prosthetic legs to remain active and lead an independent life. For most LLAs, a well-fitted prosthetic socket is the only option to interface with their prosthetic leg, however, it is a real challenge to make a prosthetic socket to interface with residual limbs accurately. One of the reasons is that there lack of accurate approaches to evaluate the pressure distribution on the residual limb accurately and effectively. To overcome this issue, the research team will develop an innovative sensing system, which permits the prosthetists to track the pressure distribution on the residual limb visually. The capability of the new sensing system will be demonstrated on lower limb amputees.

DETAILED DESCRIPTION:
A novel pressure sensing pad will be tested in the project. The purpose of these tests is to collect the safety and efficacy of the sensing pad. The research team would like to seek a Non-significant Risk claim from Institutional Review Board (IRB).

The pad will be made of materials similar to the normal liner with embedded nanotubes. The nanotubes are filled with gallium alloys, of which resistance will change based on loaded pressure. When constant current passes these tubes, the change of pressure leads to a change in temperatures around, which will excite thermal-sensitive dyes to change color. So the research team could estimate the pressure at a given area based on the color around it.

The experimental procedure includes three sets and requires 3-4 visits from each subject.

Set I procedure includes a standard socket construction, which requires 2-3 visits for the subjects to the office of a local prosthetic company. Then, a certified prosthetist will build a test socket and a customized liner to maximize the socket fit and comfort and conduct the needed alignment of the prosthetic leg. Unless it is necessary, all testing sockets will be duplications of amputees' everyday sockets.

Set II will test the accuracy of the constructed prototype on amputee subjects compared to a commercially available sensor pad, which serves as a reference. First, the research team will mount both sensing systems on the subjects. The reference sensor grid will be mounted on the residual limb directly using medical tape. After the subject dons the ENABLE sensing pad, the research team will register two sensing systems. In the end, the subjects are required to don the testing socket and walk continuously, so the measurement of the developed prototype could be stabilized. Pictures of the ENABLE will be taken and compared with the recorded pressure signals from the reference grid.

Although the reference grid and ENABLE system are designed to be put on easily, brief assistance from experimenters will be needed to ensure that the mounting procedure can be conducted appropriately.

Set III will test whether information from the ENABLE leads to appropriated socket-fit-assessments based on the response of experienced prosthetists when the prosthetists are shown the pressure distribution measured by the ENABLE under different fit conditions. All subjects will be exposed to five socket fit conditions: good and additional foam pads at four different areas shown in a random sequence. The size of the pad at each location is selected by the prosthetists based on the shape and size of the residual limbs.

Under each fitting condition, each subject will go through three trials. In each trial, the subject will walk continuously until the color of the sensing pad is stabilized. After taking high-resolution digital pictures, which cover most of the sensing area of the ENABLE, the research team will let the subject rest until the optical pattern of the ENABLE fades completely before starting a new trial.

After the experiments are finished, the subject will need to fill out a survey about the comfort of the ENABLE system. The survey will be conducted just after the experimental procedure on paper. During Set II and III, a fall prevention harness is available for the participants if it is needed. The participants are requested to self-monitor the pressure and thermal conditions on their residual limbs and encouraged to request the early termination of the experimental procedure.

ELIGIBILITY:
Inclusion Criteria:

* Unilateral transtibial amputees
* At least 1 year of experience using his/her prosthetic leg
* Has used the current socket for at least 6 months without a significant skin issue or major modification
* Can comfortably walk 3 mins without pausing to rest
* The fibula length on the residual limb must be greater than half of the length of the fibula on the unaffected side

Exclusion Criteria:

* Cognitive or visual impairment that affects the participant's ability to provide informed consent or to follow simple instructions during the experiments
* neuropathy observed on the residual limb
* regnant female

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Estimated)
Dates: Start 2021-04-20 (Actual); Primary Completion 2026-01-30 (Estimated); Study Completion 2026-02-27 (Estimated)

PRIMARY OUTCOMES:
Discomfort chart | The outcome is to evaluate the comfort of the final visit for the project (4 hours).
  Subjects are requested to fill a Wong-Baker Faces Pain Rating Scale to describe any discomfort experienced when the ENABLE system is used. This data will be used to validate that the ENABLE system is safe to use.

SECONDARY OUTCOMES:
Pressure distribution on the residual limb | The outcome is to evaluate the real pressure on the residual limb in ten 60-second walking trials.
  This outcome is measured by the developed ENABLE system and recorded by cameras after each walking trial. In three of these trials a commercially available pressure sensing pad, is also used to record the pressure distribution in the form of analog readings.

CONTACTS AND LOCATIONS:
Locations (1):
- NC State University, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
all individual participant data (IPD) that underlie results in the manuscript, which is planned to report the effectiveness of the ENABLE system.
Supporting Information: Study Protocol, ICF, CSR
Time Frame: The information will be available 6 months after the end of the experimental procedure.
Access Criteria: The statical analysis results will be available to the public with selected images collected from the experimental procedure. The full picture set will be available based on the request to the research team.

DOCUMENTS (1):
  • Informed Consent Form (2022-05-01): https://cdn.clinicaltrials.gov/large-docs/10/NCT05425810/ICF_000.pdf